CLINICAL TRIAL: NCT00407251
Title: A Phase II Study of Patupilone (EPO906A) as a Second Line Chemotherapy in Patients With Hormone Refractory Prostate Cancer
Brief Title: Study of Patupilone in Prostate Cancer Patients Who Progress After Hormone Therapy and Docetaxel Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Dr Kim Chi, British Columbia Cancer Agency
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-005/CEPO906A2402; Protocol number CEP0906A2402; OZM-005
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: refractory; prostate; hormone
MeSH Terms: interventions — epothilone B

INTERVENTIONS:
Drug: Patupilone

SUMMARY:
The purpose of this study is to determine the efficacy of patupilone chemotherapy and to find out what effects (good and bad) the drug Patupilone has on patients with prostate cancer that has progressed following hormone treatment and docetaxel chemotherapy.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer diagnosed and the second most common cause of cancer death in men in North America (Jemal 2003). Many patients with localized disease have an excellent long-term survival and high cure rates with standard approaches (D'Amico 1998). However, patients with high risk, locally advanced and metastatic disease have a poor prognosis, and although hormonal therapy in the form of medical or surgical castration can induce significant long-term remissions,development of androgen independent disease is inevitable. Androgen independent (AI) disease, also termed hormone refractory prostate cancer (HRPC), is clinically detected by a rise in prostate specific antigen (PSA) and worsening of symptoms. Once patients reach this stage, therapeutic options are limited and prognosis is poor

Patients with hormone refractory prostate cancer after docetaxel chemotherapy have limited treatment options and no treatment has been proven to be efficacious. Because of the mechanism of action and the activity of anti-microtubule agents and combinations in general for HRPC, patupilone has potential for therapeutic activity in patients with HRPC that have progressed after first line docetaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological diagnosis of adenocarcinoma of the prostate.
* Patients must have metastatic or locally recurrent disease.
* Patients must have documented evidence of PSA progression
* The PSA must be > 5 ng/mL at the time of study entry.
* ECOG performance status of 0, 1 or 2.
* Patients must have a life expectancy of at least 12 weeks in the judgment of the investigator.
* Chemotherapy: patients must have received prior docetaxel based chemotherapy (either as a single agent or in combination). Patients must have evidence of progression while receiving docetaxel based chemotherapy or within 6 months after the completion of docetaxel based chemotherapy. Prior adjuvant or neoadjuvant chemotherapy is permitted provided therapy was completed > 12 months prior to registration. Prior therapy with mitoxantrone or experimental non-cytotoxic chemotherapy is permitted (e.g. monoclonal antibodies, vaccine therapy, receptor tyrosine kinase inhibitors).
* Hormonal Therapy: Prior hormone therapy is permitted. Patients must be hormone refractory and have been previously and currently treated with androgen ablative therapy (medical or surgical castration). Therapy with LHRH agonist must continue for those prostate cancer patients already receiving this treatment at the time of enrollment. If the patient has discontinued the LHRH agonist, this must be restarted and the castrate level of testosterone must be present. Patients must have discontinued any use of non-steroidal antiandrogens (e.g. bicalutamide, nilutamide, flutamide) at least 6 weeks prior to initiation of protocol therapy.
* Radiation: Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, nonmyelosuppressive radiotherapy after consultation with the principal investigator. Prior strontium is not permitted. Patients must have had less than 30% of marrow bearing areas irradiated.
* Steroids: Current treatment with steroids are permitted provided the dose is less than or equivalent to a daily dose of prednisone of 20mg.
* Laboratory Requirements - within 7 days prior to enrollment Hematology: absolute granulocytes ≥ 1.5 x 109/Lplatelets ≥ 100 x 109/Lhemoglobin ≥ 90 g/L Biochemistry: bilirubin ≤ 1.0 x upper limit of normal serum creatinine ≤ 1.5 x upper limit of normal AST/ALT ≤ 2.5 x upper limit of normal
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre.

Exclusion Criteria:

* Patients with a history of other invasive cancer, except adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for > 3 years.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Patupilone or other agents used in the study.
* Other serious intercurrent illness of medical condition that might be aggravated by protocol treatment including: myocardial infarction within 6 months prior to study entry congestive heart failure unstable angina active cardiomyopathy unstable ventricular arrhythmia uncontrolled hypertension uncontrolled psychotic disorders serious infections active peptic ulcer disease
* HIV-positive patients receiving combination anti-retroviral therapy
* Peripheral neuropathy > grade 1.
* Patients who have received treatment with other investigational agents or anti-cancer therapy < 21 days prior to date of protocol treatment.
* Patients receiving anticoagulation with warfarin (Coumadin®).
* Patients with grade ≥ 1 diarrhea.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PSA response

SECONDARY OUTCOMES:
objective response rate
duration of response
time to PSA progression
Time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, MD, Study Chair — BC Cancer Agency - Vancouver Centre
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario